CLINICAL TRIAL: NCT01795222
Title: A Randomised Controlled Trial of Pediatric Sedation for Dental Treatment Using Oral Midazolam or Placebo
Brief Title: Midazolam Efficacy for Sedating Preschoolers Undergoing Dental Treatment
Acronym: Pedsed-I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Heloisa de Sousa Gomes, Principal Investigator, Universidade Federal de Goias
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 307/2011
Record Dates: First submitted 2012-12-19; First posted 2013-02-20 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Early Childhood Caries
Keywords: conscious sedation; stress psychological; dental care for children; child behavior; saliva
MeSH Terms: conditions — Stress, Psychological; Child Behavior | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Midazolam (Active Comparator): Midazolam oral syrup 1mg/Kg twenty minutes before starting the procedure
  Interventions: Drug: Midazolam
- placebo (Placebo Comparator): placebo oral syrup twenty minutes before starting the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midazolam — Dormire: Midazolam oral solution 2 mg/mL Sedative was administered with a syringe by the anaesthesiologist
  Other Names: Brand: Dormire (Cristalia, Sao Paulo, Brazil)
  Arms: Oral Midazolam
Drug: Placebo — Magistral formula prepared to match Dormire color and consistency, without active ingredients Placebo was administered the same way as midazolam
  Other Names: Magistral formula
  Arms: placebo

SUMMARY:
Evaluation of oral midazolam to improve children's behavior and reduces the stress and anxiety during dental treatment

DETAILED DESCRIPTION:
This study was initially planned to investigate three paediatric sedation regimens that also included the following arms:

* oral midazolam + oral ketamine + inhaled sevoflurane
* oral midazolam + oral ketamine + inhaled oxygen So, the former protocol found in the PRS registry was called PedSed-III and included the aforementioned arms.

However, there was a long delay in fund release from the funding agency (State of Goias Research Foundation - FAPEG). Although the grant was approved in the beginning of 2013, resources were released in November 2013.

We could not wait for funding release because this study was part of the MS dissertation of the principal investigator that was supposed to be concluded in the first semester of 2013. Then we decided to develop a less robust study, including only two arms: oral midazolam versus oral placebo. The other variables of the study did not change. We finished this two-arms study and have the final results for that comparison.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 5 years old, American Society of Anesthesiologists (ASA) I or II, healthy, with no cognitive impairment, presenting with early childhood caries

Exclusion Criteria:

* Children presenting with at least one of the following:
* airway obstruction and/or oral breathing;
* recent use of systemic corticosteroids
* needing less than two dental restorations;
* previous dental sedation.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
child stress | At child's awaking and arrival in the dental office, 25 min after local anesthetic administration, 25 min after dental session completion
  level of salivary cortisol according to the ELISA

SECONDARY OUTCOMES:
Child behaviour | every minute during the dental treatment up to the end of the dental session, which is estimated in 60 minutes
  child dental treatment is video recorded and then a masked observer watches the videos and categorize child behavior according to the Ohio State University Behavioral Rating Scale (OSUBRS)
sedative safety | during and twenty four hours after the procedure
  assessed according to the World SIVA adverse sedation event reporting tool

CONTACTS AND LOCATIONS:
Overall Officials: Heloisa S Gomes, DDS, Principal Investigator — Universidade Federal de Goias; Aline C Batista, PhD, Study Director — Universidade Federal de Goias
Locations (1):
- Faculty of Dentistry, Federal University of Goias, Goiânia, Goiás, Brazil